CLINICAL TRIAL: NCT04059081
Title: A Prospective Cohort of Obinutuzumab and Chlorambucil (GC) Chemotherapy for the Treatment of Elderly Patients With Chronic Lymphocytic Leukemia Including Next- Generation Sequencing (NGS)-Based Assessment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Deok-Hwan Yang (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor-Investigator, Deok-Hwan Yang, M.D., Ph.D., Chonnam National University Hospital
Organization: Chonnam National University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML40990
Record Dates: First submitted 2019-08-15; First posted 2019-08-16 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — obinutuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GC chemotherapy (Experimental): Before administration of GC chemotherapy, all patients must undergo pretreatment bone marrow biopsy. The pretreatment BM biopsy must include at least 1 long core biopsy samples and 10 cc of aspirate.
  Obinutuzumab 1000mg fixed dose will be administered intravenously (Day 1,8,15 for cycle 1 and D1 for subsequent cycles). Chlorambucil 0.5mg/kg will be administered orally (D1,15 for all cycles).
  28 days are considered as one cycle, and cycles will be repeated every 4-weeks for a total of 6 cycles.
  Interventions: Drug: Obinutuzumab

INTERVENTIONS:
Drug: Obinutuzumab — Obinutuzumab is provided as single-use vials for intravenous administration only. Obinutuzumab 1000mg fixed dose will be administered Chlorambucil would be provided as oral tablet with dose of 0.5mg/kg
  Day 1 to day 28 is considered one cycle, and cycles will be repeated every 4-weeks, until 6 cycles.

SUMMARY:
This study is prospective, open-label, single arm observational study to assess efficacy of obinutuzumab plus chlorambucil (GC) chemotherapy in treatment naïve CLL, and prognostic impact of genetic alterations for CLL using NGS.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects will be considered for inclusion in this study if they meet all of the following criteria:

  1. Newly diagnosed chronic lymphocytic leukemia
  2. Age≥ 70 years
  3. Satisfy the one of indications for starting treatment guideline

  <!-- -->

  1. Evidence of progressive marrow failure (anemia, thrombocytopenia)
  2. AIHA, thrombocytopenia refractory to steroids
  3. Massive (>6cm, LCM) or symptomatic splenomegaly
  4. Massive nodes (>10 cm) or symptomatic
  5. Progressive lymphocytosis
  6. 50% increase over 2 months or LDT < 6 months
  7. Constitutional Symptoms : weight loss > 10% in 6 months, significant fatigue, fever >38 over 2 weeks, night sweat > 1month 4. ECOG performance status 0-2 5. Total bilirubin ≤ 1.5 x ULN (upper limit of normal) 6. Aspartate aminotransferase (AST) ≤ 5 x ULN, (ALT) ≤ 5 x ULN 7. Creatinine ≤ 3.0 x ULN 8. Provide informed consent Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information

Exclusion Criteria:

1. Unmet NGS samples by bone marrow biopsy or peripheral bloods at diagnosis
2. Hairy cell leukemia or prolymphocytic leukemia
3. Uncontrolled infection
4. Therapy history with combined chemotherapy or biologic therapy prior to registration
5. History of thromboembolic episodes ≤ 3 months prior to registration
6. Active hepatitis B or C with uncontrolled disease
7. Active other malignancy requiring treatment that would interfere with the assessments of response of the lymphoma to protocol treatment
8. Any severe and/or uncontrolled medical conditions or other conditions that could adversely impact their ability to participate in the study
9. Concurrent participation in another therapeutic clinical trial.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2019-07-09 (Actual); Primary Completion 2022-07-08 (Estimated); Study Completion 2022-07-08 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 3 years
  iwCLL criteria

SECONDARY OUTCOMES:
Complete remission rate | 3 years
  No evidence of disease at the time of tumor assessment by NGS method
Progression free survival | 3 years
  the time from first dose to documented disease progression
Overall survival | 3 years
  the time from first dose to death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hallek M, Cheson BD, Catovsky D, Caligaris-Cappio F, Dighiero G, Dohner H, Hillmen P, Keating M, Montserrat E, Chiorazzi N, Stilgenbauer S, Rai KR, Byrd JC, Eichhorst B, O'Brien S, Robak T, Seymour JF, Kipps TJ. iwCLL guidelines for diagnosis, indications for treatment, response assessment, and supportive management of CLL. Blood. 2018 Jun 21;131(25):2745-2760. doi: 10.1182/blood-2017-09-806398. Epub 2018 Mar 14. PMID 29540348
- [Background] Goede V, Fischer K, Busch R, Engelke A, Eichhorst B, Wendtner CM, Chagorova T, de la Serna J, Dilhuydy MS, Illmer T, Opat S, Owen CJ, Samoylova O, Kreuzer KA, Stilgenbauer S, Dohner H, Langerak AW, Ritgen M, Kneba M, Asikanius E, Humphrey K, Wenger M, Hallek M. Obinutuzumab plus chlorambucil in patients with CLL and coexisting conditions. N Engl J Med. 2014 Mar 20;370(12):1101-10. doi: 10.1056/NEJMoa1313984. Epub 2014 Jan 8. PMID 24401022
- [Background] Fabbri G, Dalla-Favera R. The molecular pathogenesis of chronic lymphocytic leukaemia. Nat Rev Cancer. 2016 Mar;16(3):145-62. doi: 10.1038/nrc.2016.8. PMID 26911189
- [Background] Herling CD, Klaumunzer M, Rocha CK, Altmuller J, Thiele H, Bahlo J, Kluth S, Crispatzu G, Herling M, Schiller J, Engelke A, Tausch E, Dohner H, Fischer K, Goede V, Nurnberg P, Reinhardt HC, Stilgenbauer S, Hallek M, Kreuzer KA. Complex karyotypes and KRAS and POT1 mutations impact outcome in CLL after chlorambucil-based chemotherapy or chemoimmunotherapy. Blood. 2016 Jul 21;128(3):395-404. doi: 10.1182/blood-2016-01-691550. Epub 2016 May 25. PMID 27226433
- [Background] Woyach JA, Ruppert AS, Heerema NA, Zhao W, Booth AM, Ding W, Bartlett NL, Brander DM, Barr PM, Rogers KA, Parikh SA, Coutre S, Hurria A, Brown JR, Lozanski G, Blachly JS, Ozer HG, Major-Elechi B, Fruth B, Nattam S, Larson RA, Erba H, Litzow M, Owen C, Kuzma C, Abramson JS, Little RF, Smith SE, Stone RM, Mandrekar SJ, Byrd JC. Ibrutinib Regimens versus Chemoimmunotherapy in Older Patients with Untreated CLL. N Engl J Med. 2018 Dec 27;379(26):2517-2528. doi: 10.1056/NEJMoa1812836. Epub 2018 Dec 1. PMID 30501481
- [Background] Kim JA, Hwang B, Park SN, Huh S, Im K, Choi S, Chung HY, Huh J, Seo EJ, Lee JH, Bang D, Lee DS. Genomic Profile of Chronic Lymphocytic Leukemia in Korea Identified by Targeted Sequencing. PLoS One. 2016 Dec 13;11(12):e0167641. doi: 10.1371/journal.pone.0167641. eCollection 2016. PMID 27959900
- [Background] Maury S, Chevret S, Thomas X, Heim D, Leguay T, Huguet F, Chevallier P, Hunault M, Boissel N, Escoffre-Barbe M, Hess U, Vey N, Pignon JM, Braun T, Marolleau JP, Cahn JY, Chalandon Y, Lheritier V, Beldjord K, Bene MC, Ifrah N, Dombret H; for GRAALL. Rituximab in B-Lineage Adult Acute Lymphoblastic Leukemia. N Engl J Med. 2016 Sep 15;375(11):1044-53. doi: 10.1056/NEJMoa1605085. PMID 27626518
- [Background] Thomas DA, O'Brien S, Faderl S, Garcia-Manero G, Ferrajoli A, Wierda W, Ravandi F, Verstovsek S, Jorgensen JL, Bueso-Ramos C, Andreeff M, Pierce S, Garris R, Keating MJ, Cortes J, Kantarjian HM. Chemoimmunotherapy with a modified hyper-CVAD and rituximab regimen improves outcome in de novo Philadelphia chromosome-negative precursor B-lineage acute lymphoblastic leukemia. J Clin Oncol. 2010 Aug 20;28(24):3880-9. doi: 10.1200/JCO.2009.26.9456. Epub 2010 Jul 26. PMID 20660823
- [Background] Eichhorst BF, Busch R, Stilgenbauer S, Stauch M, Bergmann MA, Ritgen M, Kranzhofer N, Rohrberg R, Soling U, Burkhard O, Westermann A, Goede V, Schweighofer CD, Fischer K, Fink AM, Wendtner CM, Brittinger G, Dohner H, Emmerich B, Hallek M; German CLL Study Group (GCLLSG). First-line therapy with fludarabine compared with chlorambucil does not result in a major benefit for elderly patients with advanced chronic lymphocytic leukemia. Blood. 2009 Oct 15;114(16):3382-91. doi: 10.1182/blood-2009-02-206185. Epub 2009 Jul 15. PMID 19605849